CLINICAL TRIAL: NCT00557804
Title: Multi-Sensor Monitoring in Congestive Heart Failure Study
Brief Title: Monitoring in Congestive Heart Failure Study
Acronym: MUSIC
Status: Completed | Type: Observational
Sponsor: Corventis, Inc. (Industry)
Responsible Party: Imad Libbus, PhD, Corventis
Other Study IDs: COR-2007-001
Record Dates: First submitted 2007-11-09; First posted 2007-11-14 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MUSE clinical system — non-invasive external monitoring device

SUMMARY:
This is a multi-center, non-randomized study designed to develop an external monitor for CHF patients.

DETAILED DESCRIPTION:
Heart failure patients will be externally monitored. The collected information will be used to assess patient status.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care and heart failure clinics
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imad Libbus, PhD, Study Director — Corventis, Inc.